CLINICAL TRIAL: NCT05602857
Title: Can Training Balance, or Enjoying Music, Improve Executive Functions of Children?
Brief Title: Can Training Balance, or Enjoying Music, Improve Attention, Problem-solving and/or Behavior Control Abilities?
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Natural Sciences and Engineering Research Council, Canada (Other)
Responsible Party: Principal Investigator, Adele Diamond, professor and head of the Developmental Cognitive Neuroscience program, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: Balance and EFs study
Record Dates: First submitted 2022-10-28; First posted 2022-11-02 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2024-05

CONDITIONS: Executive Functions; Postural Balance
Keywords: executive functions; postural balance; balance training; music

STUDY DESIGN:
Intervention Model Description: Participants will be randomly allocated to one of 3 groups: Balance Training, Music Training, and business as usual (control). All groups will receive assessment of EFs and balance upon their entry into the study, 12 weeks later, and 3 months after that.
Who Masked: Participant
Masking Description: This is a single-blinded randomized controlled trial. Participants will be blinded, that is, they will not know whether we expect more EF benefit from the balance training or music condition. During recruitment we will tell the families that we are investigating whether either Balance Training (BT) and/or Music Training (MT) can improve EFs, and that we have reasons to believe that both interventions can do so. Assessment of outcomes will not be blinded, however, because the investigator (Dr. Priscilla Paz) responsible for monitoring the interventions will also be conducting the assessments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Balance Training (Experimental): Participants will follow a home-based BT intervention specifically designed by the investigators to improve postural control and balance in children. The BT program will consist of training sessions every other day (3 days a week) and a total of up to 45 minutes of balance exercises per week (15 minutes or less per session), addressing static balance (i.e., standing on one foot) and dynamic balance (i.e., balancing a book on your head while walking).
  Interventions: Other: Balance Training
- Music Training (Active Comparator): Participants will follow a home-based MT intervention designed to provide enjoyable experiences to the child participants. The sessions will occur every other day (3 days a week) for a total of up to 45 minutes per week (15 minutes or less per session) for 12 weeks. The MT program will consist of a different selection of music videos each week, including a mix of familiar and new tunes.
  Interventions: Other: Music Training
- Business as usual (No Intervention): Children assigned to this control group will follow their usual activities during the 12 weeks between initial assessment and the second assessment.

INTERVENTIONS:
Other: Balance Training — The BT program has multiple difficulty levels, and each child will progress at an individual pace tailored to their balance skills. Training sessions will emphasize top-down control of balance and contain a combination of dynamic and static balance exercises. Children and their parents will receive written step-by-step instructions, with photos, verbal and/or video instructions on their private OneDrive folder.
  To monitor compliance, whether the exercises were done properly, and evaluate a child's progress, the parent/guardian will film the sessions, and upload the video to OneDrive, so we can score the child's performance and provide them with a progress tracking chart.
  Every child will be given the equipment needed to do the balance exercises: two wooden beams that will make a 12-foot balance beam, four small wooden cubes that will raise the balance beam 5 inches off the ground, a wobble board, a hopscotch mat, one roll of painter's tape, one measuring tape, a bell, a small book.
  Other Names: Balance exercises
  Arms: Balance Training
Other: Music Training — Children assigned to MT will be asked what kind of music and what performers they like best, and what songs they like most. After those open-ended questions, they will be asked about specific songs, guided somewhat by the child's previous answers, and will watch short excerpts from music videos to see which the child would like to listen to and watch during Week 1 of the MT program. This is all to guide the selection of music videos the child will enjoy and might give some thought to.
  They will receive 10 music videos per week, through the child's private OneDrive folder, from which they can choose 4 to watch every session. Children will be instructed to not do anything else, but simply watch the videos or listen with their eyes closed.
  To monitor compliance, and to check if the child was paying attention to the music videos or just having them play in the background while doing something else, the parent/guardian will film the MT sessions, and upload the video to OneDrive.
  Other Names: enjoying music videos
  Arms: Music Training

SUMMARY:
This randomized controlled trial will investigate the hypothesis that since balance and executive functions (EFs) require a similar neural circuit and EFs are recruited when trying to maintain balance, that training balance might improve EFs as well as balance. There will be an active control condition (watching music videos) and a no-treatment condition. Children (18-12 years old) will be randomly assigned to one of these conditions for 12 weeks (36 per condition). The balance and music conditions will involve 15-min sessions 3x/week and a weekly check-in session with an investigator. Participants will be assessed pre-intervention, immediately post and 3-months post.

DETAILED DESCRIPTION:
Executive functions (EFs) are critical for success in school and in life, physical and mental health, a good quality of life, and social harmony. Indeed, EFs have even been found to be more predictive of academic & career success than socio-economic status (SES) or intelligence quotient (IQ).

It is well established that EFs depend on prefrontal cortex (PFC) and other brain regions with which it is interconnected. Recently, it has been demonstrated that much of balance (especially when there is reduced sensory input [e.g., eyes closed] or a reduced base of support [e.g., feet together or one leg raised]) requires PFC. In fact, increased PFC activity appears to compensate for sensorimotor deficits to maintain balance in older adults, and dorsolateral PFC has found to be significantly activated after external perturbation of postural stability.

It is well-established that motor learning and balance depend on the cerebellum and other interrelated brain regions. Importantly, however, the cerebellum has been shown to play an important role in EFs. The cerebellum is topographically organized in motor, cognitive and affective areas and has important anatomical connections with PFC. A growing body of recent evidence supports a close association between motor and cognitive development.

Further evidence of the close connection between EFs and motor function, especially balance, can be seen from the fact that children with impaired EFs (such as children with ADHD) tend to have impaired balance and there is an overlap between ADHD and Developmental Co-Ordination Disorder diagnosis of around 30-50%.

Further support for a close connection between balance and EFs comes from cross-sectional studies that report a positive correlation between postural stability and academic performance.

Finally, having to perform an EF task at the same time as meeting a balance challenge impairs performance on both, suggesting that they need shared neural resources.

Purpose: To see if improving balance might lead to improved EFs.

Objectives and Hypothesis Our primary objective is to determine the effect of improving postural balance, through a balance training intervention, on EFs in children 8-12 years old.

We hypothesize that training balance, especially under conditions of reduced sensory input and/or reduced base of support, will not only improve balance but also EFs. We further hypothesize that the degree of improvement in balance will be positively associated with the degree of improvement in EFs.

Although studies have supported an association between postural stability and EFs, the causal effect of balance training (without aerobic, bimanual or eye-hand coordination, and/or mindfulness components) on EFs has never been investigated. If positive results are obtained, this would be the first evidence that balance training programs might be an effective way to improve EFs. Better understanding the effect of improving balance on EFs may change our current approach to EFs training. The balance-training approach to be tried here has several advantages over traditional approaches - it can be done at home or most anywhere, a session takes only 15 minutes, it's inexpensive, it allows children to get up and move around (rather than having to stay seated at a desk), and hopefully participants will find it to be fun and enjoyable.

We wanted an active control condition that participants would expect could improve their EFs because part of the benefit from an intervention comes about just because participants expect the intervention to produce a benefit. Expectancies can become self-fulfilling prophecies so we wanted active control condition that would engender similar expectations of benefit. Watching music videos was chosen as the active control condition because of evidence that listening to music improves the cognitive functioning of adults with dementia or cognitive decline, listening to music improves mood , and improved mood leads to better EFs. We don't expect our watching-music-videos condition to improve EFs, however, because (a) children's participation is passive (they are just consumers, watching and listening) and (b) the act of watching enjoyable music videos does not place any demands on EFs (whereas doing balance exercises should).

The no-treatment group is included in case the Music Condition produces some small EF benefits, in which case the difference in benefits between the Balance and Music Conditions might not be significant. We would expect, however, that while the Balance Condition will produce EF benefits significantly greater than no-treatment, the Music Condition, if it produces EF benefits at all, will not produce ones significantly greater than no-treatment.

Study Population Assuming a significance level of 0.05, power analyses using G*Power 3.1 showed that a sample size of 30 per group would be needed to give us 80% power to detect a medium effect size (d' = 0.5) for EF change over time and for improvements in postural sway over time in children based on findings from other studies of EF or balance training in children.

Considering potential drop-out and non-compliance rates, we are allowing for 10-20% of the participants to not complete the study. Therefore, our aim is to recruit 108 participants (36 per condition).

Study Design The study interventions consist of: Balance Training (BT), Music Training (MT), and business as usual. The BT and MT interventions will run for 12 weeks, 3 sessions per week, 15 minutes each and a weekly check-in session with a member of the research staff. For the business-as-usual group, participants will have no intervention. Assessment of EFs and balance will occur at baseline, 12 weeks later, and 3 months after that.

For BT, sessions will include a combination of dynamic (i.e., balance challenges while moving, such as balancing a book on your head while walking) and static balance exercises (i.e., balance challenges while standing still, such as standing on one foot).

For MT, participants will have access to 10 music videos each week tailored to each child's specific interests from which they can choose 4 to watch in any session.

Assessments To assess the core EF skills, working memory (WM), inhibitory control (IC), and cognitive flexibility (CF), plus higher-order EF skills of problem-solving and planning, the following validated tests will be administered: N-back (WM), Re-ordering digits (WM), Hearts and Flowers (WM, IC (response inhibition), and CF), Flanker/Reverse Flanker (IC (selective attention) and CF), Stroop (IC and CF), Farmer Joe (auditory sustained attention), Tower of London (planning and problem solving), and Design Fluency (creative problem-solving). Scores for both accuracy and reaction time will be recorded.

To assess static balance, the child's center of pressure will be measured using the Wii Balance Board under the following postural stances with eyes open and eyes closed: 1) bipedal, feet shoulder-distance apart, 2) tandem, one foot in front of the other with toes of the rear foot almost touching the heel of the front foot, and 3) unipedal, standing on one leg.

To assess dynamic balance, we will measure the maximum time participants can maintain their balance standing on a wobble board with eyes open.

Statistical Analysis

First, we will look at whether variance of continuous outcome variables is normally distributed and roughly equal across conditions. Distributional characteristics of variables will be evaluated by Kolmogorov-Smirnoff goodness of fit test and by inspection of histograms. Such graphical inspection will reveal if any important deviations from normality were missed by the K-S test. Homoscedasticity will be evaluated using the Levene test. Mathematical transformations such as logarithms will be applied to improve the compliance to normality if deviations are found. In case the normality assumption is not met even after mathematical transformations, we will use the non-parametric Friedman's test as our study includes repeated outcome measures at different points in time.

We will look at whether the groups differed significantly in any background variable, like age, and whether any of these variables are significantly related to any outcome variables. We will control for any background variables that show significant effects.

To determine whether our balance training program is effective in improving balance, we will use mixed-model regression to compare participants performance on static and dynamic balance tests among all 3 groups at pre-intervention (to tell us if there were any differences among groups at the outset), post-intervention and 3-month follow-up (to tell us if any of the groups is performing significantly better than the others immediately after and/or 3 months after the intervention period). If we find a significant result, we will then do post-hoc pairwise comparisons to see which groups are significantly different from one another. Tukey or Bonferroni corrections will be used to correct for multiple comparisons potentially inflating the likelihood of finding a significant difference by chance. We will also compare degree of improvement (from pre- to post-intervention and from pre-intervention to 3-months follow-up) to see if any group(s) improved more than others and do post-hoc pairwise comparisons if any significant effects are found.

To determine whether training balance improved EFs more than enjoying music or business as usual we will again use a mixed-model regression. As described above for balance assessments, all 3 groups will be compared at pre-intervention, post-intervention and 3-month follow-up. If we find a significant result, we will then do post-hoc pairwise comparisons to see which groups are significantly different from one another. Tukey or Bonferroni corrections will be used to correct for multiple comparisons. We will also compare degree of improvement to see if any group(s) improved more than others.

To determine whether the degree of improvement in balance performance is significantly related to the degree of improvement in the EFs, we will use Pearson correlation. We will also conduct a mediation analysis using the difference in coefficients method to estimate the mediated effect of sway-area change on EF change.

ELIGIBILITY:
Inclusion Criteria

• Children between 8 to 12 years old.

Exclusion Criteria:

* Children not fluent in English
* Children with performance over the 85th percentile at screening assessment of postural balance or EFs that it leaves little room for them to improve further.
* Children taking any medication that might affect cognition (e.g., psychostimulants)
* Children undergoing EF training, which might affect their performance on EF tests.
* Children undergoing other targeted training to improve their balance (e.g., dance, yoga, tai chi, martial arts), which might affect their performance on balance tests.
* Children with severe anxiety who might find the balance training anxiety-provoking.
* Children unable to perform simple balance exercises because of a physical handicap, disability, or musculoskeletal injury.
* Children with significant hearing loss or visual impairment even with correction.
* Neither the child's parent/guardian nor other responsible person strong enough to catch the child should he or she start to fall would be available to spot the child during the weekly session in case the child is assigned to the BT intervention.

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 108 (Estimated)
Dates: Start 2023-01-25 (Actual); Primary Completion 2024-11-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in Working Memory accuracy composite score | Baseline and post-intervention (12 weeks)
  Scores for accuracy (percentage of correct responses) from each individual EF test will be analyzed separately and, using z scores, will be combined into a composite score for WM. EF tests included N-back, Re-ordering digits, hearts and flowers, flanker/reverse flanker, street test, farmer Joe, tower of London and design fluency test
Change from baseline in Inhibitory Control accuracy composite score | Baseline and post-intervention (12 weeks)
  Scores for accuracy (percentage of correct responses) from each individual EF test will be analyzed separately and, using z scores, will be combined into a composite score for IC. EF tests included N-back, Re-ordering digits, hearts and flowers, flanker/reverse flanker, street test, farmer Joe, tower of London and design fluency test
Change from baseline in Cognitive Flexibility accuracy composite score | Baseline and post-intervention (12 weeks)
  Scores for accuracy (percentage of correct responses) from each EF test will be analyzed separately and, using z scores, will be combined into a composite score for CF, and planning/problem-solving. EF tests included N-back, Re-ordering digits, hearts and flowers, flanker/reverse flanker, street test, farmer Joe, tower of London and design fluency test
Change from baseline in Planning / problem solving accuracy composite score | Baseline and post-intervention (12 weeks)
  Scores for accuracy (percentage of correct responses) from each EF test will be analyzed separately and, using z scores, will be combined into a composite score for planning/problem-solving. EF tests included N-back, Re-ordering digits, hearts and flowers, flanker/reverse flanker, street test, farmer Joe, tower of London and design fluency test
Change from baseline in Sway-area Bipedal stance, eyes closed | Baseline and post-intervention (12 weeks)
  measure os postural sway (displacements in the center of pressure (COP)) in millimetres on static bipedal stance (feet shoulder width apart) with eyes closed
Change from baseline in Sway-area Bipedal stance, eyes open | Baseline and post-intervention (12 weeks)
  measure postural sway (displacements in the center of pressure (COP)) in millimetres on static bipedal stance (feet shoulder width apart) with eyes open
Change from baseline in Sway-area Tandem stance, eyes closed | Baseline and post-intervention (12 weeks)
  measure postural sway (displacements in the center of pressure (COP)) in millimetres on static Tandem stance with eyes closed
Change from baseline in Sway-area Tandem stance, eyes open | Baseline and post-intervention (12 weeks)
  measure postural sway (displacements in the center of pressure (COP)) in millimetres on static Tandem stance with eyes open
Change from baseline in Sway-area Unipedal stance, eyes closed | Baseline and post-intervention (12 weeks)
  measure postural sway (displacements in the center of pressure (COP)) in millimetres on static Unipedal stance with eyes closed
Change from baseline in Sway-area Unipedal stance, eyes open | Baseline and post-intervention (12 weeks)
  measure postural sway (displacements in the center of pressure (COP)) in millimetres on static Unipedal stance with eyes open
Change from baseline in time standing on a wobble board, eyes open | Baseline and post-intervention (12 weeks)
  measure the maximum time participants can maintain their balance standing on a wobble board with their eyes open.

SECONDARY OUTCOMES:
Change from baseline in Working Memory accuracy composite score | Baseline and 3 months post-intervention
  Scores for accuracy (percentage of correct responses) from each individual EF test will be analyzed separately and, using z scores, will be combined into a composite score for WM. EF tests included N-back, Re-ordering digits, hearts and flowers, flanker/reverse flanker, street test, farmer Joe, tower of London and design fluency test
Change from baseline in Planning / problem solving accuracy composite score | Baseline and 3 months post-intervention
  Scores for accuracy (percentage of correct responses) from each EF test will be analyzed separately and, using z scores, will be combined into a composite score for planning/problem-solving. EF tests included N-back, Re-ordering digits, hearts and flowers, flanker/reverse flanker, street test, farmer Joe, tower of London and design fluency test
Change from baseline in Inhibitory Control accuracy composite score | Baseline and 3 months post-intervention
  Scores for accuracy (percentage of correct responses) from each individual EF test will be analyzed separately and, using z scores, will be combined into a composite score for IC. EF tests included N-back, Re-ordering digits, hearts and flowers, flanker/reverse flanker, street test, farmer Joe, tower of London and design fluency test
Change from baseline in Cognitive Flexibility accuracy composite score | Baseline and 3 months post-intervention
  Scores for accuracy (percentage of correct responses) from each EF test will be analyzed separately and, using z scores, will be combined into a composite score for CF, and planning/problem-solving. EF tests included N-back, Re-ordering digits, hearts and flowers, flanker/reverse flanker, street test, farmer Joe, tower of London and design fluency test
Change from baseline in Sway-area Bipedal stance, eyes closed | Baseline and 3 months post-intervention
  measure os postural sway (displacements in the center of pressure (COP)) in millimetres on static bipedal stance (feet shoulder width apart) with eyes closed
Change from baseline in Sway-area Bipedal stance, eyes open | Baseline and 3 months post-intervention
  measure os postural sway (displacements in the center of pressure (COP)) in millimetres on static bipedal stance (feet shoulder width apart) with eyes closed
Change from baseline in Sway-area Tandem stance, eyes closed | Baseline and 3 months post-intervention
  measure postural sway (displacements in the center of pressure (COP)) in millimetres on static Tandem stance with eyes closed
Change from baseline in Sway-area Tandem stance, eyes open | Baseline and 3 months post-intervention
  measure postural sway (displacements in the center of pressure (COP)) in millimetres on static Tandem stance with eyes closed
Change from baseline in Sway-area Unipedal stance, eyes closed | Baseline and 3 months post-intervention
  measure postural sway (displacements in the center of pressure (COP)) in millimetres on static Unipedal stance with eyes closed
Change from baseline in Sway-area Unipedal stance, eyes open | Baseline and 3 months post-intervention
  measure postural sway (displacements in the center of pressure (COP)) in millimetres on static Unipedal stance with eyes closed
Change from baseline in time standing on a wobble board, eyes open | Baseline and 3 months post-intervention
  measure the maximum time participants can maintain their balance standing on a wobble board with their eyes open.

CONTACTS AND LOCATIONS:
Overall Officials: Adele Diamond, PhD, Principal Investigator — University of British Columbia
Locations (1):
- Developmental Cognitive Neuroscience Lab, Department of Psychiatry, UBC, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No